CLINICAL TRIAL: NCT04636346
Title: Evaluation of Compass: A Group Clinical Program in Psycho-Oncology Using Acceptance and Commitment Therapy to Address Fear of Recurrence/Progression in Cancer Survivors
Brief Title: COMPASS: A Group ACT Program for Cancer Patients Treated at UCSF
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 19805
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Cancer
Keywords: Survivorship
MeSH Terms: conditions — Neoplasms | interventions — Acceptance and Commitment Therapy; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COMPASS (Psychoeducational / Behavioral Program): Group Acceptance and Commitment Therapy program as part of clinical service for cancer patients
  Interventions: Behavioral: Acceptance and Commitment Therapy; Other: Questionnaires

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Seven group sessions
Other: Questionnaires — Outcomes measured include anxiety, depression, fear of recurrence, psychological flexibility, mindfulness; values based living, and quality of life. Participants completed surveys at 4 time points, pre and post, and two follow-up time points.

SUMMARY:
Cancer Center Psychosocial services (Psycho-Oncology) offers group psychoeducational and behavioral programs as part of its clinical service for cancer patients and services at the Helen Diller Family Comprehensive Cancer Center. Clinical outcomes and acceptability/feasibility and implementation process data from these programs are routinely gathered in an effort to engage in continuous quality improvement for the department.

DETAILED DESCRIPTION:
For this project, the study team is proposing to retrospectively analyze a de-identified data set of these data to report on pilot data on preliminary outcomes, acceptability and feasibility of the implementation of the COMPASS: Acting Mindfully for a Valued Life, based upon Acceptance and Commitment Therapy, an evidence-based behavioral intervention and facilitated by a licensed clinical psychologist in our department. This intervention was implemented as a series of clinical offerings for seven 7-session groups between September 2015 and October 2018 for 113 individual cancer patients and survivors. Outcomes measured include anxiety, depression, fear of recurrence, psychological flexibility, mindfulness; values based living, and quality of life. Participants completed surveys at 4 time points, pre and post, and two followup time points. Measures of demographics, satisfaction and feasibility/acceptability were also collected. Insights gathered from this study will be used to inform articles, grant applications and conference presentations on the implementation of behavioral interventions for cancer patients and survivors.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Treated for any kind of cancer at University of California, San Francisco
* Sufficient cognitive ability to participate in group activities as determined by their attending medical oncologist or surgeon

Exclusion Criteria:

* Non-English speaking
* Treated elsewhere for cancer
* Psychiatric illness that would affect the ability to participate in a group activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied will include the participants of the COMPASS Program offered by the Cancer Center Psychosocial services (Psycho-Oncology) that consented to having their responses for the surveys to be used for research purposes. The participants of COMPASS were adult cancer patients across different cancer types. Participants that had previously consented to having their responses to the surveys kept for research purposes will have their responses accessed and kept as a part of a de-identified data set. No direct subject contact will be included
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Changes in the Patient Reported Outcome Measurement Information System (PROMIS) Anxiety Short Form scores over time | Up to 1 year
  The PROMIS Anxiety Short form consists of 2 items addressing patient anxiety with item response scores ranging from 1 (never) to 5 (Always). Raw scores are converted to scaled T-scores with higher scores indicating a greater level of anxiety. Significant changes over time and trends in patient reported outcomes will be analyzed via student's T-test.
Changes in the Patient Reported Outcome Measurement Information System (PROMIS) Depression Short Form scores over time | Up to 1 year
  The PROMIS Depression Short form consists of 4 items addressing patient depression with item response scores ranging from 1 (never) to 5 (Always). Raw scores are converted to scaled T-scores with higher scores indicating a greater level of depression. Significant changes over time and trends in patient reported outcomes will be analyzed via student's T-test.
Changes in Acceptance and Action Questionnaire II (AAQ-II) scores over time | Up to 1 year
  The AAQ-II is a 7 item questionnaire used to track how participants are doing with applying psychological flexibility skills in their daily life. Item scores range from 1 ("never true") to 7 ("always true":), and total scores are computed by adding up responses for each question. Higher total scores mean less flexibility, while lower total scores mean more flexibility.
Changes in the Functional Assessment of Cancer Therapy scale (FACT-G) scores over time | Up to 1 year
  The FACT-G is a 27-item questionnaire designed to measure four domains of health related quality of life (HRQOL) in cancer patients with 4 domains of interest: Physical, social, emotional, and functional well-being. Each tem response score ranges from 0 (not at all) to 5 (very much). The total score is a sum of the subscale scores, with a range from 0 - 108. The higher the score, the better the HRQOL.
Changes in the Valuing Questionnaire (VQ) scores over time | Up to 1 year
  The VQ is a 10-item scale designed to measure how consistently an individual has been living with their self-determined values and is helpful when administered during a course of Acceptance and Commitment Therapy (ACT). Two subscale scores are measured: Progress and Obstruction. Progress items (Range = 0 to 30) are defined as enactment and perseverance in living consistently with one's values. Higher scores represent a closer alignment between one's internal values and one's actions. Obstruction (Range = 0 to 30) represents the extent to which various disruptions "got in the way" of valued living. Higher scores represent more interference with living consistently with one's values. Total scores are calculated by summing the raw scores and calculating percentile ranks. When used as a monitoring tool during a course of ACT, successful treatment is indicated by increasing Progress Scores and decreasing Obstruction Scores.
Changes in The Fear of Cancer Recurrence Index (FCRI) severity subscale scores over time | Up to 1 year
  The nine-item FCRI evaluates the presence and severity of intrusive thoughts associated with FCR. Each item is rated on a Likert scale ranging from 0 ("not at all" or "never") to 4 ("a great deal' or "all the time"). A higher score indicates higher levels of FCR.
Changes in the Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being (FACIT-SP-12) scores over time | Up to 1 year
  The FACIT-SP-12 is a 12 item questionnaire which measures a participants spiritual well-being for the past 7 days. Item responses range from 0 (not at all) to 4 (very much). The sum of the item scores are used to calculate a total FACIT-SP-12 score ranging from 0 to 48. The higher the score, the better the QOL/spiritual well-being.
Changes in Five Facet Mindfulness Questionnaire (FFMQ) scores over time | Up to 1 year
  The FFMQ is a 39-item questionnaire that measures five factors which represent elements of mindfulness. The five facets are Observing, Describing, Acting with awareness, Non-judging of inner experience, and Non-reactivity to inner experience. Item scores range from 1 ("never or very rarely true") to 5 ("very often or always true":), and total scores are computed by adding up responses for the questions that fall into each facet, for a range of 8-40 per facet with the exception of the Non-react scores which range from 7-35. Higher scores on the Observe, React, and Non-react facets indicate higher levels of mindfulness and higher scores on the Act with Awareness and Non-judge items indicate less mindfulness.
Changes in Happiness Index Profile (HI/P10) scores over time | Up to 1 year
  The HI/P10 is a 10-item questionnaire assessing positive affect, intention, and resiliency. Each item is scored from 0 (strongly disagree) to 10 (strongly agree). HI/P10 scores are calculated by adding the scores for each item to generate a total score out of 100.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Chesney, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No